CLINICAL TRIAL: NCT03797547
Title: Real Life Study in Myopic Neovascularization
Acronym: VIC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: VIC
Record Dates: First submitted 2018-08-28; First posted 2019-01-09 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Myopic Choroidal Neovascularisation
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: AFLIBERCEPT — Patients will be treated following a real life protocol and according to the French recommendation

SUMMARY:
This is a multi centre, single arm, prospective observational phase 4 study in naive or pretreated patients with myopic neovascularization. The patients will be treated with intravitreal injections of Aflibercept following a real life protocol.

This sudy aims to evaluate the visual acuity during a 36 months period of time.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged 18 years and more under reliable method of contraception for woman with childbearing potenteial (hormonal or any intrauterine devices).
* High myopy defined by refractive error ≤ -6 D or History of high myopia among pseudophakic patient or patient treated with refractive surgery
* Patient with active CNVm
* • Patients naïve or Patients pretreated with previous history of laser photocoagulation or PDT or by other anti-VEGF treatments who did not receive injection since the last 3 month

  * with OCT or angiography examination

Exclusion Criteria:

* Treatment with an anti VEGF administrated by intravitreal injection within 1 months prior to baseline in the study eye.
* Treatment with PDT or laser administrated within 6 months prior to baseline in the study eye.
* History of vitrectomy in the study eye
* History of any other retinal disease
* VA less than 20/250

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Active mCNV among:
  * Naïve patients.
  * Patients with previous history of laser photocoagulation or PDT, with no history of anti-VEGF.
  * Patients with previous history of other anti-VEGF treatments.including ranibizumab or bevacizumab, with sustaining mCNV activity, who did not receive injection since the last 3 month
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
visual acuity measurement | 6, 12, 24 and 36 months
  Efficacy measurement will be performed by mean change of "ETDRS" for Best Corrected Visual Acuity evaluation (ETDRS score at 4 meters) from baseline to 6, 12, 24 and 36 month after initation of treatment by aflibercept

SECONDARY OUTCOMES:
visual acuity measurement in naive patient | 12, 24 and 36 months
  Efficacy measurement will be performed by mean change of "ETDRS" for Best corrected visual acuity evaluation from baseline to month 12, 24 and 36 after initation of treatment by aflibercept in naïve patients
visual acuity measurement after other treatment such as laser, pdt visudyneor other IVT treatment | 6, 12, 24 and 36 months
  Efficacy measurement will be evaluated by mean change of "ETDRS" for Best corrected visual Acuity evaluation after initation of treatment by aflibercept after switch from other treatment such as laser, visudyne PDT or other IVT treatment, after 6, 12, 24 and 36 months of treatment with Eylea
pourcentage of patients who gain more than or equal of 15 letters | 6,12,24 and 36 months
  Efficacy measurement will be evaluated by pourcentage of patients who gain more than or equal of 15 letters at 6, 12, 24 and 36 months after initiation of treatment with aflibercept within naïve or after switch from other treatment such as laser, visudyne PDT or other IVT treatment,
Anatomics parameters by oct | 6, 12, 24 and 36 months
  Evaluation of anatomic parameters will be perfomed after 6,12, and 24 and 36 months of treatment with Eylea based on OCT parameters :
  On SD-OCT :
  Distance from CNV lesion to the fovea measured on the scan joining the fovea to the foveal edge of the mCNV Exudation assessed by presence of intraretinal cysts or subretinal fluid Central retinal thickness
Anatomics parameters by color photographs | 6, 12, 24 and 36 months
  On color retinal photographs:
  Presence of retinal hemorrhage Presence of macular atrophy or lacquer cracks,
Anatomic parameters by fluoresceine angiography or angiography oct | 6, 12, 24 and 36 months
  On fluoresceine angiography if deemed necessary by the investigator : diffusion during late phases On angiography OCT : neovascular network visualisation

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Poitiers, Poitiers, France